CLINICAL TRIAL: NCT03406429
Title: Pilot Study of Repetitive Transcranial Magnetic Stimulation in Patients With Primary Progressive Aphasia.
Brief Title: rTMS as a Treatment for PPA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Mark C. Eldaief, MD, Assistant Professor of Neurology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017P002319
Record Dates: First submitted 2017-12-20; First posted 2018-01-23 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Logopenic Variant Primary Progressive Aphasia; Non-Fluent Primary Progressive Aphasia
Keywords: rTMS; PPA
MeSH Terms: conditions — Primary Progressive Nonfluent Aphasia

STUDY DESIGN:
Intervention Model Description: Within-subject crossover design
Masking Description: Through use of SHAM rTMS stimulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- PPA patients (Experimental): All study participants will carry a diagnosis of Primary Progressive Aphasia (PPA), either the logopenic or the non-fluent variant. All participants will receive the same study interventions in a within-subject crossover design.
  Interventions: Device: Active rTMS; Device: SHAM rTMS

INTERVENTIONS:
Device: Active rTMS — All study participants will receive one block of active rTMS. Each block will consist of daily sessions of 20Hz active rTMS delivered to the left dorsolateral prefrontal cortex (dlPFC) over five days (Monday through Friday).
Device: SHAM rTMS — All study participants will receive one block of SHAM rTMS. Each block will consist of daily sessions of 20Hz SHAM rTMS delivered to the left dorsolateral prefrontal cortex (dlPFC) over five days (Monday through Friday).

SUMMARY:
Primary progressive aphasia (PPA) includes three variants. Two such variants, the non-fluent/agrammatic variant (nfvPPA) and the logopenic variant (lvPPA), are characterized by progressive word-finding difficulties and effortful speech. Efforts to slow or halt this progression have been largely unsuccessful. As such, there is a desperate need for novel treatment strategies in PPA.

Repetitive transcranial magnetic stimulation (rTMS) is a safe, non-invasive way of stimulating cortical targets in a focal and reproducible manner. Therapeutic benefits from rTMS have been demonstrated when it is applied in many sequential sessions. For example, repeated sessions of rTMS to left dorsolateral prefrontal cortex (dlPFC) is approved by the US Food and Drug administration as a treatment for major depressive disorder. With respect to language, high frequency rTMS increases the response rate for picture naming in healthy individuals. rTMS has also been shown to improve the number of correct naming responses in patients with Alzheimer's disease. Further, in a sham controlled study, Cotelli and colleagues demonstrated that in a group of 10 nfvPPA patients high frequency rTMS over the left and right dlPFC during object and action naming tasks improved the percent of correct responses for action, but not object naming. Finally, in a sham controlled single case study, Finocchiaro et al. applied high frequency rTMS to the left inferior mid-frontal gyrus for 3 sessions consisting of five consecutive days (treatment or sham). They found a significant and lasting improvement in the patient's performance on verb production when comparing active rTMS to sham rTMS or baseline. These studies have contributed valuable insights into the potential use of rTMS in treating the language symptoms of PPA patients.

DETAILED DESCRIPTION:
15-20 patients with a confirmed diagnosis of either nfvPPA or lvPPA (made by a specialized clinician) will be recruited. Patients must have a mild to moderate language impairment and must be native English speakers. Exclusion criteria include contraindications to receiving Magnetic Resonance Imaging (MRI) scanning or rTMS (e.g. metallic or electromagnetically activated implants, cranial mass lesions, surgical aneurysm clips), the presence of significant medical, neurological or psychiatric co-morbid symptoms and patients without study partners.

It will take approximately 2 weeks to complete this research study, but the exact timing will vary according to patient, investigator and equipment availability. Each patient will have a total of up to 11 study visits. Greater than 11 visits may take place in the event that patients' language improves significantly following rTMS in order to test the sustainability of the improvement. Visits will take place at the MGH Martinos Center for Biomedical Imaging.

The first visit (lasting 3-4 hours) will include obtainment of informed consent, baseline assessments, and a baseline MRI scan (which will be used for subsequent rTMS targeting). After this, patients will return for two blocks of 20Hz rTMS to left dlpfc: one in which they receive active rTMS and one in which they receive sham rTMS. Both active and sham rTMS will be delivered as high frequency stimulation (20 hertz, 20Hz). To accomplish this, an rTMS coil capable of delivering active or sham stimulation will be employed. Order of active and sham blocks will be counterbalanced across participants. During each block rTMS (active or sham) will be administered daily for 5 days (Monday through Friday). Neuropsychological testing, including thorough language evaluations, will be done before and after each block of rTMS. Repeat MRI imaging will be performed at the end of each of the two blocks. rTMS visit durations will be as follows: Monday visits will last approximately 3-4 hours, Tuesday, Wednesday and Thursday visits will last approximately 1-2 hours and Friday visits will last approximately 5 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, age 18-90, who carry a diagnosis of either the logopenic (lvPPA) or agrammatic non-fluent (nfvPPA) variants of Primary Progressive Aphasia (PPA). Patients must have been observed for at least one year by a specialized clinician.
2. Patients must have at least mild to moderate language impairment.
3. Patients must be native English speakers.
4. Patients must have a study partner (e.g. spouse, sibling or adult child) who can accompany them to every study visit.

Exclusion Criteria:

1. Any history of seizures, unexplained loss of consciousness or a first-degree family member with epilepsy.
2. Any history of significant co-occurring neurological illness unrelated to neurodegeneration associated with PPA (e.g. multiple sclerosis), or significant medical problems (e.g. poorly controlled diabetes/hypertension or cancer within 5 years).
3. Active symptoms of major depressive disorder, bipolar disorder, schizophrenia, substance use disorder or significant premorbid intellectual disability according to Diagnostic Statistical Manual (DSM-5) criteria.
4. Magnetic Resonance Imaging (MRI) evidence of significant cerebrovascular disease, hydrocephalus or the presence of a space-occupying intra-cranial mass.
5. Contraindications to MRI or repetitive transcranial magnetic stimulation (rTMS) including: cardiac pacemaker or pacemaker wires, neurostimulators, implanted pumps, metal in the body (rods, plates, screws, shrapnel, dentures, intrauterine device), surgical aneurysm clips in the head, previous neurosurgery or cochlear implants.
6. In line with published Massachusetts General Hospital (MGH) Institutional Review Board (IRB) guidelines for rTMS, pregnancy must be ruled out by urine ß-Human Chorionic Gonadotropin if answers to screening questions suggest that pregnancy is possible and if female participants are premenopausal and of child-bearing age. Subjects will not be able to enroll if they are breastfeeding.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Language Assessment Battery | At the beginning and end of each rTMS block.
  This will include tests of speech production, confrontation naming, sentence completion.
MRI Imaging | At the baseline visit and at the end of each rTMS block.
  This will include observed changes in resting-state functional connectivity and cortical thickness occurring as a result of the stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finocchiaro C, Maimone M, Brighina F, Piccoli T, Giglia G, Fierro B. A case study of Primary Progressive Aphasia: improvement on verbs after rTMS treatment. Neurocase. 2006 Dec;12(6):317-21. doi: 10.1080/13554790601126203. PMID 17182394
- [Background] Cotelli M, Manenti R, Petesi M, Brambilla M, Cosseddu M, Zanetti O, Miniussi C, Padovani A, Borroni B. Treatment of primary progressive aphasias by transcranial direct current stimulation combined with language training. J Alzheimers Dis. 2014;39(4):799-808. doi: 10.3233/JAD-131427. PMID 24296814